CLINICAL TRIAL: NCT01950026
Title: Temperature Skin Check in Different Ethnic Groups After Cryotherapy Application
Brief Title: Temperature Skin Check After Cryotherapy Application
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Mauricio Correa Lima, expert, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125.608
Record Dates: First submitted 2013-07-03; First posted 2013-09-25 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Body Temperature Changes
Keywords: skin temperature; ethnic groups; cryotherapy
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- white (Experimental): cryotherapy application
  Interventions: Procedure: cryotherapy application
- black (Experimental): cryotherapy application
  Interventions: Procedure: cryotherapy application
- Brown (Experimental): cryotherapy application
  Interventions: Procedure: cryotherapy application
- asian (Experimental): cryotherapy application
  Interventions: Procedure: cryotherapy application

INTERVENTIONS:
Procedure: cryotherapy application — * Height, weight and BMI verification
  * subjects in supine position after 20 minutes of resting
  * cryotherapy application by cold thermal bag (thermoGel brand) size P
  * 15-20 cm above the ASIS
  * temperature verified before and after cryotherapy application with an infrared thermometer CA 380 CASON brand, Brazil

SUMMARY:
The aim of this study was to reheat the skin in different ethnic groups after application of cryotherapy.

DETAILED DESCRIPTION:
It is a clinical randomized cross-sectional. This study was approved by the Ethics Committee of the Universidade Paulista - UNIP under protocol number 125 608 of 18/10/2012.

The study included 24 subjects randomly recruited from both sexes and from four different ethnic groups: white, brown, black and asian with different ages, individuals intolerant to cold, suffering any change in skin sensitivity, illness from infectious diseases or previously diagnosed to respond negatively to the use of cold were excluded.

The survey was conducted in the clinic Physiotherapy Universidade Paulista - UNIP in light and airy ambience, with recording of the mean daily temperature in degrees Celsius planned for the capital of São Paulo by newsletter Climatempo available and accessed http://www.climatempo.com.br/previsao-do-tempo/cidade/ Before all applications, the average temperature obtained in the days from the application was 21.93° Celsius.

For obtaining of personal data and anthropometric evaluations, a data sheet prepared by the authors to self-fulfillment, and then calculated the BMI of subjects, if in doubt, check the height and body mass was performed before the application of cryotherapy. Participants were divided into 4 groups of different ethnicities - white, brown, black and asian; ethnicity was proven through the birth certificates of volunteers, according to the classification described by the Brazilian Institute of Geography and Statistics - IBGE.

All participants were maintained in supine position for 20 minutes to rest and stabilization of body temperature, sleep after receiving an application through the cold thermal bag Thermo Gel ® brand size "P" consisting of a cellulose-based gel for subsequently receiving of cryotherapy in the middle third of the right thigh and left earlier, leaving 15-20 cm from the anterior superior iliac spine - ASIS side tested, depending on the stature of the individual being assessed and 5 cm away from the surface to be evaluated, according to manufacturer's instructions. The temperature was verified on site described before, during and after applications of cryotherapy which lasted for 30 minutes and then recorded. To check the temperature after application of cryotherapy was used a thermometer brand CASON ® INFRARED THERMOMETER AC 380 (- 32 º C 380 º C).

ELIGIBILITY:
Inclusion Criteria:

* belong to ethnic groups requested

Exclusion Criteria:

* suffering any change in skin sensitivity, illness of an infectious nature or previously diagnosed diseases that respond negatively to the use of cold

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
changes in skin cooling | two months
  It was verified skin temperature of the subject in the supine position with them prior to the application of cryotherapy during application (at 3, 5, 10, 15, 20, 25 min) and after the application retitrada ice and after 30 minutes of implementation. Measurements were obtained in degrees Celsius with an infrared thermometer brand CASON Model CA380 recorded in a collection daos elaborated by authors

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio C Lima, expert, Principal Investigator — Paulista University
Locations (1):
- Rehabilitation Center of Universidade Paulista, São Paulo, São Paulo, Brazil